CLINICAL TRIAL: NCT01171859
Title: A Single Center, Twelve-month, Open-label, Prospective Study Followed by a Six-month Withdrawal Period to Evaluate the Efficacy, Tolerability, Safety and Pharmacokinetics of Doxycycline in Combination With Tauroursodeoxycholic Acid in Transthyretin Amyloidosis
Brief Title: Safety, Efficacy and Pharmacokinetics of Doxycycline Plus Tauroursodeoxycholic Acid in Transthyretin Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giampaolo Merlini, Prof., Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOXYTUDCA2010; 2010-020422-17 (EudraCT Number)
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Transthyretin Amyloidosis
Keywords: amyloidosis; transthyretin; doxycycline; Tauroursodeoxycholic acid
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — Doxycycline; ursodoxicoltaurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxycycline + Tauroursodeoxycholic acid (Experimental)
  Interventions: Drug: Doxycycline + Tauroursodeoxycholic acid

INTERVENTIONS:
Drug: Doxycycline + Tauroursodeoxycholic acid — doxycycline 100 mg twice a day for 12 months; tauroursodeoxycholic acid 250 mg three times a day for 12 months

SUMMARY:
This study is being conducted to explore the potential benefits of a twelve-month doxycycline (at the best tolerated dose of 200 mg/day) and tauroursodeoxycholic acid (750 mg/day) treatment on disease progression in patients affected by transthyretin amyloidosis, including: 1) patients not eligible for liver transplantation; 2) patients eligible for liver transplantation, as a "bridge" therapy between the time of diagnosis and surgery, with the aim of stabilizing the disease; 3) patients showing disease progression after liver transplantation performed since at least 1 year.

It is a phase II, therapeutic exploratory, two-part, 18-month, single centre, prospective study.

Part I is a 12-month, open label treatment period in which doxycycline (200 mg/day, continuously) and tauroursodeoxycholic acid (750 mg/day continuously) are administered to 40 consenting subjects with transthyretin amyloidosis. Part II is a withdrawal period in which subjects will be monitored for disease progression. During part I, subjects will be evaluated at baseline (study Day 0), and then after 3, 6, 9 and 12 months of doxycycline plus tauroursodeoxycholic acid treatment or at premature treatment discontinuation; during part II, they will be assessed at months 15 and 18. Monthly phone contacts and blood tests will be performed to monitor potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens;
* Molecular definition of the transthyretin (TTR) mutation or immunohistochemical staining of amyloid fibrils with anti-TTR antibody;
* ECOG performance status (PS) 0, 1, 2;
* New York Heart Association (NYHA) class ≤III
* Systolic blood pressure ≥100 mmHg (standing)
* Must have symptomatic organ involvement with amyloid to justify therapy; must have evidence of neuropathy and/or cardiomyopathy progression after liver transplantation performed since at least one year.
* Contraception for women of childbearing potential. Medically approved contraception could include abstinence. A negative serum pregnancy test is required prior to initiation of treatment with study medication.

Exclusion Criteria:

* Liver transplantation in the previous 12 months or liver transplantation anticipated in less than 6 months;
* ALT and/or AST ≥ 2 x Upper Normal Limit (UNL);
* Alkaline phosphatase ≥ 2 x UNL;
* Creatinine clearance < 30 ml/min;
* Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study;
* Echocardiographic ejection fraction < 50%;
* Other neuropathies, due to vitamin B12 deficiency, alcoholism, hypothyroidism, uremia, diabetes mellitus, vasculitides;
* History of poor compliance;
* History of hypersensitivity to any of the ingredients of the study therapies;
* Use of any investigational drug, device (or biologic) within 4 weeks prior to study entry or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Response rate to doxycycline + tauroursodeoxycholic acid treatment | One year
  A responder is a subject with:
  * a modified body mass index (mBMI) reduction of less than 10% and a change in the Neurologic Impairment Score-Lower Limbs (NIS-LL) <2 (in subjects with peripheral neuropathy);
  * a modified body mass index (mBMI) reduction of less than 10% and an increase in N-terminal natriuretic peptide type B (NT-proBNP) concentration of less than 30% or < 300 pg/mL (in subjects with isolated cardiomyopathy).

SECONDARY OUTCOMES:
Number of patients experiencing treatment-emergent adverse events | One year
Change in quality of life | Every six months
  SF-36 scale
doxycycline pharmacokinetics (PK) | Every three months
response in autonomic dysfunction, sensory-motor peripheral neuropathy and visceral organ involvement | One year
  response assessed according to the Kumamoto Scale score
neurologic response | One year
  response assessed by motor and sensory nerves conduction studies
Incidence of patients discontinuing from the study because of clinical or laboratory adverse events | One year

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Merlini, MD, Principal Investigator — IRCCS Policlinico San Matteo
Locations (1):
- Amyloid Research and Treatment Centre, Biotechnology Research Laboratories, Pavia, Pavia, Italy

REFERENCES:
- [Background] Cardoso I, Saraiva MJ. Doxycycline disrupts transthyretin amyloid: evidence from studies in a FAP transgenic mice model. FASEB J. 2006 Feb;20(2):234-9. doi: 10.1096/fj.05-4509com. PMID 16449795
- [Background] Macedo B, Batista AR, Ferreira N, Almeida MR, Saraiva MJ. Anti-apoptotic treatment reduces transthyretin deposition in a transgenic mouse model of Familial Amyloidotic Polyneuropathy. Biochim Biophys Acta. 2008 Sep;1782(9):517-22. doi: 10.1016/j.bbadis.2008.05.005. Epub 2008 Jun 3. PMID 18572024
- [Background] Cardoso I, Martins D, Ribeiro T, Merlini G, Saraiva MJ. Synergy of combined doxycycline/TUDCA treatment in lowering Transthyretin deposition and associated biomarkers: studies in FAP mouse models. J Transl Med. 2010 Jul 30;8:74. doi: 10.1186/1479-5876-8-74. PMID 20673327